CLINICAL TRIAL: NCT03430128
Title: Perioperative Immunonutrition for Patients Undergoing Cytoreductive Surgery (CRS) and Hyperthermic Intraperitoneal Chemotherapy
Brief Title: Perioperative Immunonutrition for Patients Undergoing CRS and HIPEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2016/3063
Record Dates: First submitted 2018-01-30; First posted 2018-02-12 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Peritoneal Metastases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators and the clinical team which manages the patient, will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral IMPACT (Experimental): Perioperative immunonutrition will commence 5-7 days prior to surgery, and will continue for 5-7 days post-surgery, as soon as the patient is able to consume full feeds as instructed by his/her primary physician.
  The recommended dose for IMPACT immunotherapy is one packet, to be taken three times a day.
  Interventions: Dietary Supplement: IMPACT immunotherapy
- Standard Nutrition (ENSURE) (Active Comparator): Standard nutritional supplementation will commence 5-7 days prior to surgery, and will continue for 5-7 days post-surgery, as soon as the patient is able to consume full feeds as instructed by his/her primary physician.
  Interventions: Dietary Supplement: ENSURE

INTERVENTIONS:
Dietary Supplement: IMPACT immunotherapy — Powdered formula that is pre-packaged in individual packets which the patients will be instructed to mix with water before consumption.
  Arms: Oral IMPACT
Dietary Supplement: ENSURE — Liquid milk formula available over the counter
  Arms: Standard Nutrition (ENSURE)

SUMMARY:
Patients with peritoneal disease commonly present with symptoms of abdominal distension and subacute intestinal obstruction. This results in poor oral intake leading to these patients often presenting in a malnourished state.

CRS and HIPEC can potential provide improve survival for these patients, however can be a hazardous procedure, involving multi-organ resections. The risk is especially high in poorly nourished patients.

The study investigators hypothesize that perioperative immunonutrition can reduce wound infections and length of hospital stay, and improve perioperative outcomes. To the investigators' knowledge, it has not been evaluated in patients undergoing CRS and HIPEC.

ELIGIBILITY:
Inclusion Criteria:

1. All patients planned for CRS and HIPEC, with sufficient time (5 to 7 days) prior to surgery for start of nutritional supplements are eligible
2. All patients must be able to provide informed consent
3. There are no restrictions to use of contraception

Exclusion Criteria:

1. Patients who are not able to provide informed consent will be excluded.
2. Patients with a diagnosis of diabetes mellitus will be excluded.
3. Patients not fit for surgery or those who undergo surgery under emergency situations will be excluded.
4. Patients who have intestinal obstruction and not able to consume the nutritional supplements orally will be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-23 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Baseline wound infection rates | From date of surgery to date that wound is healed, up to 30 days from surgery

SECONDARY OUTCOMES:
Peri-operative complications | Within 30 days from surgery
Length of stay | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Teo, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No